CLINICAL TRIAL: NCT04037189
Title: Treatment of Leukemia and Lymphoma in Children With Ataxia Telangiectasia- A Retrospective Study
Brief Title: Treatment of Leukemia and Lymphoma in Children With Ataxia Telangiectasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Israeli Society for Pediatric Hematology-Oncology (Other); International BFM Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: 0132-19-RMC
Record Dates: First submitted 2019-07-21; First posted 2019-07-30 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-08

CONDITIONS: Ataxia Telangiectasia; Leukemia; Lymphoma
MeSH Terms: conditions — Ataxia Telangiectasia; Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ataxia telangiectasia (A-T) is a multisystem disease with diverse manifestations, including progressive neurodegeneration, immunodeficiency, respiratory disease, and genomic instability. One of the most important features of A-T is the increased predisposition to cancer, especially to lymphoid malignancies. Patients with A-T are generally excluded from collaborative clinical trials, their treatment outcomes and toxicity profiles have rarely been reported, and little is currently known concerning the treatment intensity required to provide a reasonable balance between efficacy and toxicity. The aims of this study are to build a large international de-identified database of children with A-T treated for leukemia and lymphoma, to investigate epidemiology and outcome of treatment, toxicity profiles and risk factors which impact outcome, in order to eventually enable the generation of data-based treatment recommendations for this population.

DETAILED DESCRIPTION:
Ataxia telangiectasia (A-T) is a multisystem disease with diverse manifestations, including progressive neurodegeneration, immunodeficiency, respiratory disease, and genomic instability. A-T is caused by biallelic mutations in the ATM gene, a major activator of the cellular response to DNA double strand breaks. One of the most important features of A-T is the increased predisposition to cancer. Lymphoid malignancies represent the majority of cancers. The treatment of cancer in children with A-T is extremely challenging, due to severe co-morbidities and a significantly increased risk of cancer therapy-related toxicities. Patients with A-T are generally excluded from collaborative clinical trials, their treatment outcomes and toxicity profiles have rarely been reported, and little is currently known concerning the treatment intensity required to provide a reasonable balance between efficacy and toxicity. The optimal treatment approach is controversial; some advocate treatment by standard chemotherapeutic protocols, while others advise initial protocol modifications with chemotherapy dose reductions. Due to the rarity of this disorder, there is an unmet need for an international collaboration for data collection concerning treatment, toxicity and outcome in children with cancer and A-T. Data will be collected from patient files, including patient characteristics and history, AT manifestations, malignancy characteristics, treatment, chemotherapy doses, treatment response, toxicity and outcome.

The aims of the study are to build a large international de-identified database of children with A-T treated for leukemia and lymphoma, to investigate epidemiology and outcome of treatment, toxicity profiles and risk factors which impact outcome, in order to eventually enable the generation of data-based treatment recommendations for this population.

This study will not involve the use of specimens or participant contact. All the data required have already been collected during the treatment of the participants, and is available in patient records.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with ataxia telangiectasia and leukemia or lymphoma
* Age 0-21

Exclusion Criteria:

-Age greater than 21 years

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults diagnosed with ataxia telangiectasia and leukemia or lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-07-28 (Actual); Primary Completion 2021-10-28 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 5 years
  Assess 5 and 3-year event-free survival
Overall survival | 5 years
  Assess 5 and 3-year overall survival
Cumulative incidence of relapse | 5 years
  Assess 5-year cumulative incidence of leukemia/lymphoma relapse
Cumulative incidence of treatment-related mortality | 2 years
  Assess 2-year cumulative incidence of treatment-related mortality
Cumulative incidence of second malignancies | 5 years
  Assess 5-year cumulative incidence of second malignancies

SECONDARY OUTCOMES:
Cause and timing of death | 5 years
  Determine cause of death and timing of death in relation to specific elements of leukemia/lymphoma therapy (by questionnaire)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Elitzur, MD, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel